CLINICAL TRIAL: NCT01184677
Title: Comparison of the Size 3 ProsealTM Laryngeal Mask Airway Versus Size 4 in Anaesthetized, Non-paralyzed Women: A Randomised Controlled Trial
Brief Title: ProSeal Laryngeal Mask Airway (LMA) Size 3 vs 4 in Non-paralyzed Female Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kim Mihyun, professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: ProSeal LMA 3 vs 4
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Oropharyngeal Injury
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group size 4 (Placebo Comparator)
  Interventions: Device: insertion of the PLMA
- Group size 3 (Experimental): ProSeal LMA size 3 is inserted to the patients of Group size 3.
  Interventions: Device: insertion of the ProSeal LMA (PLMA)

INTERVENTIONS:
Device: insertion of the ProSeal LMA (PLMA) — ProSeal LMA size 3 is inserted to the patients of Group size 3.
  Other Names: insertion; ProSeal LMA size 3
  Arms: Group size 3
Device: insertion of the PLMA — ProSeal LMA size 4 is inserted to the patients of Group size 4.
  Other Names: insertion; ProSeal LMA size 4
  Arms: Group size 4

SUMMARY:
The investigators hypothesize that ProSeal laryngeal mask airway (PLMA) of smaller size would reduce the incidence of mucosal injury.

DETAILED DESCRIPTION:
The ProSealTM laryngeal mask airway (PLMA; Laryngeal Mask Co. Limited, Mahe, Seychelles) is a laryngeal mask device with an added dorsal cuff to improve the seal and a drainage tube to prevent aspiration and gastric insufflations(Brain, Verghese et al. 2000).Despite its utility, there are complications associated with PLMA insertion such as sore throat and mucosal injury including oropharyngeal blood.

The purpose of this randomized controlled study is to determine if size 3 PLMA would induce less mucosal damage indicated by blood on the cuff than size 4 in non-paralyzed female patients. The secondary objective of this study is to compare insertion time, number of attempts, oropharyngeal leak pressure, hemodynamic variables, and incidence of complications with size 3 and 4 PLMA.

ELIGIBILITY:
Inclusion Criteria:

* female
* aged 18-80 yr
* American Society of Anesthesiologists physical status Ⅰ-Ⅱ
* scheduled to undergo short outpatient gynecological procedures using ProSealTM LMA (PLMA) for anesthesia

Exclusion Criteria:

* a known or predicted difficult airway
* recent sore throat
* mouth opening less than 2.5 cm
* body mass index > 35 kg/m2
* at risk of aspiration.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
blood on the ProSeal LMA | from the start of ProSeal LMA insertion until the end of the anesthesia (around 30min , mostly less than 60min)
  The incidence of blood on the proseal LMA upon removal of the device is assessed in each group.

SECONDARY OUTCOMES:
hemodynamic variables | from induction of anesthesia until immediately after the Proseal LMA insertion
  mean arterial pressure and heart rate before and after the Proseal LMA insertion are measured.
insertion time | from grasping the Proseal LMA until an effective airway is established
seal pressure | after successful insertion of Proseal LMA
  oropharyngeal leak pressure
other intraoperative complications | from successful insertion of PLMA until the end of the anesthesia
  airway leak, failed ventilation, regurgitation/aspiration, laryngospasm, cough/gag/retching/hiccup.
postoperative complications | from removal of Proseal LMA until discharge from recovery room
  sore throat and hoarseness

CONTACTS AND LOCATIONS:
Overall Officials: Mihyun Kim, professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea